CLINICAL TRIAL: NCT06773377
Title: Study of the Prognostic Impact of CD44 on Renal Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wafaa Ashraf Fawzy, Doctor, Assiut University
Other Study IDs: CD44 on Renal Cell Carcinoma
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. Study the expression of CD44 in various histopathological types of RCC.
2. Study the association between CD44 expression and other clinicopathological parameters
3. study the impact of CD44 expressions in tumor and patients' survival

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is the seventh most common form of neoplasm in the developed world, accounting for approximately 2% of global cancer diagnoses and deaths and increase in burden worldwide [1]. RCC is a rising worldwide incidence estimated at 400 000 new cases annually, and a worldwide mortality rate approaching 175 000 deaths per year [2].

RCC mortality rate is 2-3% per decade, therefore novel therapies directed against RCC are needed. At the same time despite advancements in diagnostic techniques, up to 30% of newly diagnosed patients already present with metastases, and a large portion of patients that undergo surgical treatment experience the RCC recurrence, therefore drugs targeted against metastasis initiating cells would be of great interest in the future [3].

The major risk factors for RCC, including smoking, obesity, hypertension , occupational exposure to harmful substances and chronic kidney disease must be taken in consideration [4, 5] The WHO 2022 Classification of Urinary and Male Genital Tumors (5th edition) is molecular-driven and contains major revisions compared to the earlier classification from 2016. The fourth edition divided renal tumors into four major broad categories: clear cell renal tumors, papillary renal cell tumors, oncocytic and chromophobe renal tumors, and collecting duct tumors [6]. Novel entities included in the WHO 2022 classification are eosinophilic solid and cystic renal cell carcinoma (ESC RCC), anaplastic lymphoma kinase (ALK)-rearranged RCC and ELOC (formerly TCEB1)-mutated RCC [7].

The most consistent prognostic factors are tumor size, stage, grade, and histopathological parameters such; tumor necrosis, histological types, microvascular invasion [5, 8].

To date, the only potential curative treatment is surgery. However, 20-30% of patients with RCC develop local or distal recurrence within years of a nephrectomy [9]. The recurrence of RCC after surgery is a major factor that affects negatively the patient survival. On the other hand, multiple unfavorable prognostic factors such as perineal fat invasion, tumor size, size of the largest involved lymph node and extra-nodal extension are neither reliable nor accurate enough for predicting the therapeutic response [10].

Recent studies have shown that several molecular and genetic biomarkers could play a role in predicting response to therapy [11].

Cancer stem cells (CSCs) together with cancer aggressiveness, including treatment resistance such as chemo/radiotherapy, and targeted treatment are responsible not only for cancer development, but also for disease recurrence, progression and metastatic spread [3].

CD44 is one of CSCs and a cell membrane glycoprotein involved in diverse cellular processes including cell motility, proliferation, apoptosis, and angiogenesis, when there is a pathologic change, become characteristic of malignancy [12].

Unsurprisingly, CD44 is expressed in many cancers, including those of the skin, blood, head and neck, lung, breast, stomach, colon, prostate, uterus, and brain. CD44 is overexpressed on cancer stem cells, and its expression in various cancers has provided an ample opportunity for the treatment of patients with chemoresistance malignancy [13].

Some studies explained that high expression of CD44 in RCC was associated with metastasis, poor prognosis [14]. CD44 expression turned out to be a promising target as it is involved in the regulation of cell proliferation, differentiation and apoptosis induction [15].

In our study we will assess the expression of CD44 in various histopathological types of RCC. understanding their biology is mandatory to define novel potential prognostic and therapeutic targets for all RCC subtypes.

ELIGIBILITY:
Inclusion Criteria:

* patient must be more than 18 years
* Patients with complete pathological data

Exclusion Criteria:

* The presence of any other organ malignancies
* Patients who lost follow-up after nephrectomy less than 3-year,
* Patients with incomplete pathological data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with RCC who had undergone radical or partial nephrectomy, between 2014 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Study of the prognostic impact of CD44 on renal cell carcinoma. | Baseline
  assess the expression of CD44 in various histopathological types of RCC. understanding their biology is mandatory to define novel potential prognostic and therapeutic targets for all RCC subtypes.